CLINICAL TRIAL: NCT05975281
Title: Comparison of Neuropathic Pain Symptoms in Hand Osteoarthritis and Rheumatoid Arthritis
Brief Title: Neuropathic Pain Symptoms in Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Department of Physical Medicine and Rehabilitation, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 28052023
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Neuropathic Pain
Keywords: hand osteoarthritis; neuropathic pain; neuropathic symptom; rheumatoid arthritis
MeSH Terms: conditions — Neuralgia; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hand osteoarthritis: Those diagnosed with hand osteoarthritis according to the American College of Rheumatology (ACR) criteria
- Rheumatoid arthritis: Those diagnosed with rheumatoid arthritis according to the American College of Rheumatology (ACR) criteria

SUMMARY:
It was aimed to compare neuropathic pain symptoms in hand osteoarthritis and rheumatoid arthritis.

DETAILED DESCRIPTION:
The patients with hand osteoarthritis or neuropathic complaints accompanying rheumatoid arthritis who applied to the Physical Medicine and Rehabilitation Clinic of our hospital will be included. In both patient groups, the duration, character and treatments of their complaints will be compared. Neuropathic pain will be evaluated with the Visual Analog Score (VAS), Dolor Neuropathic 4 Questions (DN-4) and Pain Detect pain questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Hand Osteoarthritis and Rheumatoid Arthritis
* Presence of neuropathic complaints

Exclusion Criteria:

* History of hand injury, peripheral nerve injury, fracture, and hand operation in the last 3 months
* Do not want to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with hand osteoarthritis or neuropathic complaints accompanying rheumatoid arthritis who applied to the Physical Medicine and Rehabilitation Clinic of Şişli Hamidiye Etfal Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-27 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Day 1
  0-10 ; higher score : severe pain
DN-4 | Day 1
  0-10 ; > 4 neuropathic pain
Pain detect pain questionnaire | Day 1
  0-38 ; < 13 negative, 13-18 unclear, >18 positive

CONTACTS AND LOCATIONS:
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)